CLINICAL TRIAL: NCT04068779
Title: Long-term Clinical Outcomes in Patients With FFR GuidEd-DeFERred CoRonAry Lesions, Assessed by IVUS Analysis
Acronym: REFERRAL
Status: Completed | Type: Observational
Sponsor: Keimyung University Dongsan Medical Center (Other)
Responsible Party: Principal Investigator, Yun-kyeong Cho, professor, Keimyung University Dongsan Medical Center
Other Study IDs: 2019-05-048
Record Dates: First submitted 2019-08-23; First posted 2019-08-28 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-02

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study was a multicenter retrospective study that included intravascular ultrasound (IVUS) in patients with delayed stent insertion based on fractional flow reserve (FFR) in moderately narrowed coronary lesions. We would like to see the effect of lesion characteristics on clinical course.

DETAILED DESCRIPTION:
From January 2007 to August 2014, patients who meet the criteria for selection and exclusion from Keimyung University Dongsan Hospital, Seoul National University Hospital, Inje University Busan Paik Hospital, and Ulsan University Hospital are included.

1. Target patient screening The database will select patients who meet the selection and exclusion criteria.
2. target patient characteristics The age, sex, smoking status, medical history (hypertension, diabetes mellitus, hyperlipidemia), diagnosis, and left ventricular blood count measured by echocardiography should be checked through a computerized medical record.
3. coronary angiography Coronary angiography images of the subjects in the blinded state are analyzed to investigate the length of lesions, reference vessel diameter, and minimal vessel diameter.
4. intravascular ultrasound In the blinded state, the vessel's vessel area, plaque area, lumen area, etc. are measured by analyzing intravascular ultrasound images of the patient using EchoPlaque (Indec Systems, Mountain View, CA).

ELIGIBILITY:
Inclusion Criteria:

* Subject over 19 years old
* Patients with mild or moderate stenosis lesions on coronary angiography
* Patients with lesions with FFR values greater than 0.80
* Patients with analytical intravascular ultrasound images

Exclusion Criteria:

* Left main lesion
* History of coronary artery bypass grafting
* Patients with lower left ventricular ejection fraction (<25%)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From January 2007 to August 2014, patients who meet the criteria for selection and exclusion from Keimyung University Dongsan Hospital, Seoul National University Hospital, Inje University Busan Paik Hospital, and Ulsan University Hospital are included.
Sampling Method: Probability Sample
Enrollment: 459 (Actual)
Dates: Start 2019-05-31 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
patient-oriented composite outcome | during 5-year
  all-cause death, myocardial infarction and any revascularization

CONTACTS AND LOCATIONS:
Locations (1):
- KeimyungUniversity, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: No